CLINICAL TRIAL: NCT07387185
Title: Development and Validation of an Artificial Intelligence System for Detection and Characterization of Small Bowel Mucosal Atrophy in Celiac Disease and Non-Celiac Enteropathies: A Multicenter Observational Study
Brief Title: AI System for Detection and Characterization of Chronic Enteropathies
Status: Recruiting | Type: Observational
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Collaborators: Fondazione IRCCS Policlinico San Matteo, Pavia, Italy (Unknown); Ospedale Valduce, Como (Unknown); Azienda Ospedale Università Padova, Padova (Unknown); IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other); ASST Cremona, Cremona (Unknown); Azienda Ospedaliero-Universitaria Città della Salute e della Scienza di Torino (Unknown); Fondazione Poliambulanza Istituto Ospedaliero, Brescia (Unknown); ASST degli Spedali Civili di Brescia , Brescia (Unknown); IRCCS Policlinico San Donato, Milano (Unknown); Azienda Socio-Sanitaria Territoriale (ASST) di Pavia (Unknown); Azienda Unità Sanitaria Locale della Romagna, Ravenna (Unknown); ASST Lecco, Lecco (Unknown); Fondazione IRCCS Ca' Granda Ospedale Maggiore Policinico, Milano (Unknown); Academic Unit of Gastroenterology, Sheffield Teaching Hospitals, Sheffield, UK (Unknown)
Responsible Party: Sponsor
Other Study IDs: CTSPV36-24
Record Dates: First submitted 2026-01-28; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Celiac Disease; Small Bowel Mucosal Atrophy or Lesions; Non-celiac Enteropathies
Keywords: Artificial Intelligence; Endoscopy; Deep Learning; Computer-Aided Diagnosis; Small Bowel
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Enteropathy Cohort (CD/NCE): Adult patients (>=18 years) with suspected or confirmed Celiac Disease or Non-Celiac Enteropathies undergoing small bowel endoscopy.
- Control Cohort: Adult patients (>=18 years) undergoing small bowel endoscopy who do not have enteropathy or other small bowel pathological lesions (negative controls).
- Other Small Bowel Lesion Cohort: Adult patients (>=18 years) undergoing small bowel endoscopy who who do not have Celiac Disease or Non-Celiac Enteropathies but have other small bowel pathological lesions.

SUMMARY:
Coeliac disease (CD) is an immune-mediated enteropathy leading to small intestinal mucosal atrophy. Diagnosis relies on serology and duodenal biopsies, but it can be complicated by patchy lesions and differential diagnosis with Non-Celiac Enteropathies (NCEs). This multicenter observational study aims to develop and validate an Artificial Intelligence (AI) system to detect and characterize small bowel mucosal atrophy and other pathological findings using endoscopic imaging. The study involves a retrospective phase for training the AI model and a prospective phase to validate its diagnostic accuracy compared to standard human assessment.

DETAILED DESCRIPTION:
The study is a multicenter observational non-profit study with a total expected duration of 36 months. It aims to address the challenges in diagnosing CD and NCEs, specifically the subjective nature of endoscopic evaluation and inter-observer variability.

The study proceeds in two phases:

1. Model Development (Retrospective): Training of Deep Learning algorithms on anonymized endoscopic images/videos to identify mucosal atrophy and other lesions (e.g., angiodysplasia, ulcers, polyps).
2. Validation (Prospective): Enrolling patients undergoing small bowel endoscopy to validate the AI system's performance.

The system aims to provide analysis to assist endoscopists, reducing missed lesions and improving diagnostic accuracy.

Validation of the AI system will be performed offline on recorded anonymized endoscopy videos collected prospectively during the validation phase.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age ≥18 years).
* Patients undergoing endoscopic investigation of the small bowel (endoscopy or capsule endoscopy)

Exclusion Criteria:

* Inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing endoscopic investigation of the small bowel (endoscopy or capsule endoscopy) for suspected or known celiac disease, non-celiac enteropathies or other small bowel conditions
Sampling Method: Probability Sample
Enrollment: 380 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Performance of the AI System | Through study completion (36 months)
  Evaluation of Accuracy, Sensitivity, and Specificity of the AI system in detecting intestinal mucosal atrophy and other major pathological findings compared to the gold standard (histology/expert consensus).

SECONDARY OUTCOMES:
Comparison of Diagnostic Performance (No AI-assistance vs AI-assisted) | Through study completion (36 months)
  Comparison of accuracy, sensitivity, and specificity of gastroenterologists performing assessment with and without the assistance of the AI system.
Inter-observer Agreement | Through study completion (36 months)
  Measurement of agreement between the AI system and expert gastroenterologists in evaluating the extent of mucosal atrophy.

CONTACTS AND LOCATIONS:
Locations (1):
- ICS Maugeri IRCCS, Pavia, PV, Italy

IPD SHARING:
Plan to Share IPD: Undecided